CLINICAL TRIAL: NCT02944448
Title: A Randomized, Double-Blind, Placebo-Controlled, Titration-to-Effect Study of Orally Administered CR845 in Patients With Osteoarthritis of the Hip or Knee
Brief Title: A Study Evaluating Pain Relief and Safety of Orally Administered CR845 in Patients With Osteoarthritis of Hip or Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-CLIN2002-PO
Record Dates: First submitted 2016-10-04; First posted 2016-10-25 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
Keywords: Osteoarthritis; Hip; Knee; CR845; Analgesic; Kappa opioid; difelikefalin
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CR845 tablet 1 mg (Active Comparator): Dosing twice a day (BID) for a total of 8 weeks, with each dose administered at least 2 hours prior to or after a meal.
  Interventions: Drug: CR845 tablet 1 mg
- CR845 tablet 2.5 mg (Active Comparator): Dosing twice a day (BID) for a total of 8 weeks, with each dose administered at least 2 hours prior to or after a meal.
  Interventions: Drug: CR845 tablet 2.5 mg
- CR845 tablet 5 mg (Active Comparator): Dosing twice a day (BID) for a total of 8 weeks, with each dose administered at least 2 hours prior to or after a meal.
  Interventions: Drug: CR845 tablet 5 mg
- Placebo tablet (Placebo Comparator): Dosing twice a day (BID) for a total of 8 weeks, with each dose administered at least 2 hours prior to or after a meal.
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: CR845 tablet 1 mg — CR845 tablets will be provided as 1 mg enteric-coated tablets. All tablets are white in color with no markings and are identical in appearance, regardless of dose and treatment.
  Arms: CR845 tablet 1 mg
Drug: CR845 tablet 2.5 mg — CR845 tablets will be provided as 2.5 mg enteric-coated tablets. All tablets are white in color with no markings and are identical in appearance, regardless of dose and treatment.
  Arms: CR845 tablet 2.5 mg
Drug: CR845 tablet 5 mg — CR845 tablets will be provided as 5 mg enteric-coated tablets. All tablets are white in color with no markings and are identical in appearance, regardless of dose and treatment.
  Arms: CR845 tablet 5 mg
Drug: Placebo tablet — Placebo tablets will be provided as enteric-coated tablets. All tablets are white in color with no markings and are identical in appearance, regardless of dose and treatment.
  Arms: Placebo tablet

SUMMARY:
The study schedule consists of a Screening Period (up to 14 days), a blinded 4- week Titration-to-Effect Period with weekly visits, a blinded 4-week Maintenance Treatment Period at the optimal dose level determined for each patient, and a 1-week Follow-up Period.

Eligible patients will be randomized to receive either CR845 or placebo in a 2:1 ratio. Every patient will be started on a 1-mg dose of CR845 or matching placebo. During the post-randomization Titration-to-Effect period, the dose of study drug may be increased to 2.5 mg or 5 mg in a double-blind fashion. Patients may know their dose is being changed but will not know whether they were randomization to active study drug or placebo. Approximately 330 patients will be enrolled in this study.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, titration-to-effect study of orally administered CR845 in patients with osteoarthritis of the hip or knee.

The study schedule consists of a Screening Period (up to 14 days), a blinded 4- week Titration-to-Effect Period with weekly visits, a blinded 4-week Maintenance Treatment Period at the optimal dose level determined for each patient, and a 1-week Follow-up Period.

Eligible patients will be randomized to receive either CR845 or placebo in a 2:1 ratio. Randomization will be stratified based on a patient's primary OA joint (knee vs. hip). Every patient will be started on a 1-mg dose of CR845 or matching placebo. During the post-randomization Titration-to-Effect period, the dose of study drug may be increased to 2.5 mg or 5 mg in a double-blind fashion.

Patients may know their dose is being changed but will not know whether they were randomized to active study drug or placebo. Approximately 330 patients will be enrolled in this study.

During the Screening, Titration-to-Effect and Follow-up Period, pain intensity scores will be obtained at specified time points. Blood sampling and safety assessments will be conducted during this period as well.

The use of rescue medication for the treatment of any pain (including but not limited to headache, menstrual cramps, or non-target joint pain) during the study will be discussed with the patients at the Screening Visit. Acetaminophen is the only allowable rescue medication for pain beginning from Day -5 until the end of the Maintenance Treatment Period. Starting at the Screening Visit Acetaminophen will be provided as 325-mg tablets and its use (number of tablets taken in the previous 24 hours) will be reported each evening in the patient diary.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provides written informed consent to participate in the study prior to any study procedures.
2. Is able to speak, read, and communicate clearly in English or Spanish; is able to understand the study procedures.
3. Male or female ≥ 25 years of age.
4. Body mass index (BMI) ≤ 40 kg/m2.
5. Has OA of the hip or knee according to American College of Rheumatology (ACR) criteria.
6. Reports an average pain intensity level ≥ 5 in the index joint at Screening on a 0-10 NRS scale.
7. Is either opioid-naïve (defined as taking < 10 mg a day of morphine equivalent 14 days prior to screening) or opioid-experienced. If receiving opioid analgesic medication for OA, patients must be on a stable dose ≤ 40 mg of morphine equivalents for 14 days prior to screening.
8. Willing to discontinue currently used pain medications beginning 5 days prior to the Baseline Visit and throughout the study. Acetaminophen use is allowed. (Section 8.8)
9. If female:

   1. Of childbearing potential - the patient must be willing to practice an acceptable form of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives, or abstinence from sexual intercourse) for the duration of treatment and for at least 3 days following the last dose of study drug.
   2. Of non-childbearing potential - the patient must be surgically or biologically sterile (hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or postmenopausal for at least 1 year).
10. If male, the patient must be surgically or biologically sterile. If not sterile, the patient must agree to use an acceptable form of birth control with a heterosexual partner (as described in inclusion criterion #9) or abstain from sexual relations during the treatment period and for 3 days following the last dose of study drug.
11. Is free of other physical, mental, or medical conditions that, in the opinion of the Investigator, would make study participation inadvisable.
12. Reports a daily pain intensity score in the index joint ≥ 5 (on a 0-10 NRS scale) during 4 or more of the last 7 days prior to randomization, with 2 consecutive days ≥ 5 occurring just prior to randomization

Exclusion Criteria:

Inclusion Criteria:

A patient will be eligible for enrollment if the following criteria are met:

1. Voluntarily provides written informed consent to participate in the study prior to any study procedures.
2. Is able to speak, read, and communicate clearly in English or Spanish; is able to understand the study procedures.
3. Male or female ≥ 25 years of age.
4. Body mass index (BMI) ≤ 40 kg/m2.
5. Has OA of the hip or knee according to American College of Rheumatology (ACR) criteria.
6. Reports an average pain intensity level ≥ 5 in the index joint at Screening on a 0-10 NRS scale.
7. Is either opioid-naïve (defined as taking < 10 mg a day of morphine equivalent 14 days prior to screening) or opioid-experienced. If receiving opioid analgesic medication for OA, patients must be on a stable dose ≤ 40 mg of morphine equivalents for 14 days prior to screening.
8. Willing to discontinue currently used pain medications beginning 5 days prior to the Baseline Visit and throughout the study. Acetaminophen use is allowed. (Section 8.8)
9. If female:

   1. Of childbearing potential - the patient must be willing to practice an acceptable form of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives, or abstinence from sexual intercourse) for the duration of treatment and for at least 3 days following the last dose of study drug.
   2. Of non-childbearing potential - the patient must be surgically or biologically sterile (hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or postmenopausal for at least 1 year).
10. If male, the patient must be surgically or biologically sterile. If not sterile, the patient must agree to use an acceptable form of birth control with a heterosexual partner (as described in inclusion criterion #9) or abstain from sexual relations during the treatment period and for 3 days following the last dose of study drug.
11. Is free of other physical, mental, or medical conditions that, in the opinion of the Investigator, would make study participation inadvisable.
12. Reports a daily pain intensity score in the index joint ≥ 5 (on a 0-10 NRS scale) during 4 or more of the last 7 days prior to randomization, with 2 consecutive days ≥ 5 occurring just prior to randomization

Exclusion Criteria:

1. Has had a joint replacement in the index joint.
2. Has received an intra-articular injection of corticosteroids or hyaluronic acid in the index joint within 3 months prior to the Screening Visit.
3. Has started a new medication for chronic illness within 30 days prior to the Screening Visit.
4. Is receiving opioid analgesic treatment for OA of the hip or knee at a dose > 40 mg of morphine equivalent.
5. Uses antipsychotics, antiepileptics, sedatives, hypnotics, or antianxiety agents, selective serotonin reuptake inhibitors (SSRIs), tricyclic antidepressants with a dose change <30 days prior to day 1 of the study.
6. Has a history or current diagnosis of substance dependence (except caffeine or nicotine) or alcohol abuse, according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
7. Has a positive urine drug screen for drugs of abuse at Screening.
8. Has been diagnosed with a condition of hyperhidrosis (excessive sweating) or primary hypodipsia (a reduced sense of thirst).
9. Has a history (within 6 months) of clinically meaningful orthostatic changes in vital signs OR, at Screening, has a decrease in systolic blood pressure by > 20 mm Hg or a decrease in diastolic blood pressure by 10 mm Hg together with an increase in heart rate of > 30 beats per minute when transitioning from supine to standing measurements.
10. Has a medical condition (e.g., a cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine [adrenal hyperplasia], immunologic, dermatologic, neurologic, oncologic, or psychiatric) or a significant laboratory abnormality that, in the Investigator's opinion, would jeopardize the safety of the patient or is likely to confound the study measurements.
11. Has had any gastric bypass surgery (for weight loss).
12. Has a corrected QT interval of >450 msec in males, >470 msec in females, or clinically significant abnormality on screening ECG.
13. Has a serum sodium level > 143 mmol/L at Screening.
14. Has impaired renal function indicated by serum creatinine > 2 × the reference upper limit of normal (ULN).
15. Has a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × the reference ULN, or total bilirubin > 2 × the ULN at Screening.
16. Has, in the opinion of the Investigator, any clinical signs of dehydration or hypovolemia (e.g., symptomatic hypotension) or associated laboratory abnormalities (e.g., elevated hematocrit or elevated blood urea nitrogen [BUN] > 1.5 × the reference ULN) at Screening.
17. Has taken opioid or non-opioid pain medication (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs] such as naproxen or cyclooxygenase-2 inhibitors) within 5 days prior to study drug administration. Acetaminophen use is allowed. (Section 8.8)
18. Has received another investigational drug within 30 days prior to Baseline or has planned to participate in another clinical trial while enrolled in this study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Stauffer, DO, MBA, Study Director — Cara Therapeutics
Locations (32):
- United States (32):
  - Cara Therapeutics Study Site, Birmingham, Alabama
  - Cara Therapeutics Study Site, Peoria, Arizona
  - Cara Therapeutics Study Site, Phoenix, Arizona
  - Cara Therapeutics Study Site, Carmichael, California
  - Cara Therapeutics Study Site, San Diego, California
  - Cara Therapeutics Study Site, Tustin, California
  - Cara Therapeutics Study Site, Homestead, Florida
  - Cara Therapeutics Study Site, Jupiter, Florida
  - Cara Therapeutics Study Site, Lake Worth, Florida
  - Cara Therapeutics Study Site, Miami, Florida
  - Cara Therapeutics Study Site, Oldsmar, Florida
  - Cara Therapeutics Study Site, Orlando, Florida
  - Cara Therapeutics Study Site, Plantation, Florida
  - Cara Therapeutics Study Site, South Miami, Florida
  - Cara Therapeutics Study Site, Tampa, Florida
  - Cara Therapeutics Study Site, Savannah, Georgia
  - Cara Therapeutics Study Site, Hazelwood, Missouri
  - Cara Therapeutics Study Site, Omaha, Nebraska
  - Cara Therapeutics Study Site, Las Vegas, Nevada
  - Cara Therapeutics Study Site, Berlin, New Jersey
  - Cara Therapeutics Study Site, Binghamton, New York
  - Cara Therapeutics Study Site, Rochester, New York
  - Cara Therapeutics Study Site, Cincinnati, Ohio
  - Cara Therapeutics Study Site, Oklahoma City, Oklahoma
  - Cara Therapeutics Study Site, Duncansville, Pennsylvania
  - Cara Therapeutics Study Site, Charleston, South Carolina
  - Cara Therapeutics Study Site, Greenville, South Carolina
  - Cara Therapeutics Study Site, Austin, Texas
  - Cara Therapeutics Study Site, Dallas, Texas
  - Cara Therapeutics Study Site, Plano, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- CR845 Tablet: Every patient was started on a twice daily (BID) 1 mg dose of CR845. During the post-randomization Titration-to-Effect Period, the dose of study drug may have been increased to 2.5 mg BID or 5 mg BID in a double-blind fashion.
- Placebo Tablet: Twice daily dosing (BID)
Period: Overall Study
Arm/Group | CR845 Tablet | Placebo Tablet
Started | 316 | 160
Completed | 227 | 136
Not Completed | 89 | 24
Not completed — Adverse Event | 37 | 6
Not completed — Lack of Efficacy | 8 | 5
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 25 | 7
Not completed — Withdrawal by Subject | 14 | 4
Not completed — Sponsor did not supply drug in time | 0 | 1
Not completed — Noncompliant with dosing | 1 | 0
Not completed — Abnormal laboratory values | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CR845 Tablet | Placebo Tablet | Total
Number analyzed (Participants) | 316 | 160 | 476
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.26) | 60.8 (10.26) | 60.5 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 89 | 299
  Male | 106 | 71 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 61 | 33 | 94
  White | 245 | 122 | 367
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 8 With Respect to the Weekly Mean of the Daily 24-hour Pain Intensity for the Index Joint as Measured by the Numeric Rating Scale (NRS).
Description: 11-point NRS scale where 0 = no pain, and 10= pain as bad as you can imagine
Time Frame: Baseline, Week 8
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- CR845 Tablet: Dosing twice a day (BID) for a total of 8 weeks, with each dose administered at least 2 hours prior to or after a meal.
  During the post-randomization Titration-to-Effect Period, the dose of study drug may have been increased to 2.5 mg BID or 5 mg BID in a double-blind fashion.
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 316 | 160
score on a scale | -2.3 (0.14) | -2.4 (0.19)
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.7093, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.5]

2. Secondary Outcome: Change From Baseline in the Western Ontario & McMaster Osteoarthritis (WOMAC) Index Total Score at Week 8
Description: The WOMAC Index is a self-administered assessment used to measure pain, stiffness, and physical function in patients with osteoarthritis. The WOMAC Index contains 24 questions across 3 different sub-scales (pain, stiffness, and function) all with scoring 0-10 (0 = No Pain/Stiffness/Difficulty, 10 = Extreme Pain/Stiffness/Difficulty). Each WOMAC Index Subscale score (Pain/Stiffness/Function) is calculated as the sum of all scores within that subscale. The pain subscale consists of five scores from 0-10, 0 is no pain 10 is extreme pain possible for a range of 0 - 50 points. The stiffness subscale consists of two scores from 0-10, 0 is no stiffness 10 is extreme stiffness possible for a range of 0 - 20 points. The function subscale consists of 17 scores from 0-10, 0 is no difficulty and 10 is extreme difficulty, for a range of 0 - 170 points. The WOMAC Index Total Score is calculated as the sum of all 24 scores (range of 0-240).
Time Frame: Baseline, Week 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 223 | 133
score on a scale | -62.4 (3.28) | -59.7 (4.34)
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.6007, Mixed Models Analysis; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-13.1 to 7.6]

3. Secondary Outcome: Change From Baseline in the WOMAC Pain Intensity Sub-scale Score at Week 8
Description: The pain subscale consists of five scores from 0-10, 0 is no pain 10 is extreme pain possible for a range of 0 - 50 points.
Time Frame: Baseline, Week 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 223 | 133
score on a scale | -13.5 (0.70) | -12.7 (0.92)
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.4563, Mixed Models Analysis; Median Difference (Final Values) = -0.8, 95% CI 2-sided [-3.0 to 1.4]

4. Secondary Outcome: Change From Baseline in the WOMAC Stiffness Sub-scale Score at Week 8
Description: The stiffness subscale consists of two scores from 0-10, 0 is no stiffness 10 is extreme stiffness possible for a range of 0 - 20 points.
Time Frame: Baseline, Week 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 223 | 133
score on a scale | -5.7 (0.29) | -5.6 (0.38)
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.8693, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.0 to 0.8]

5. Secondary Outcome: Change From Baseline in the WOMAC Function Sub-scale Score at Week 8
Description: The function subscale consists of 17 scores from 0-10, 0 is no difficulty and 10 is extreme difficulty, for a range of 0 - 170 points.
Time Frame: Baseline, Week 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 223 | 133
score on a scale | -43.1 (2.34) | -41.5 (3.10)
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.6516, Mixed Models Analysis; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-9.1 to 5.7]

6. Secondary Outcome: Proportion of Patients With at Least 30% Improvement From Baseline in the Weekly Mean Pain Intensity at Week 8
Description: A patient's pain response to treatment is defined as the percent improvement from baseline with respect to the weekly mean of "average pain in the last 24 hours" pain score during the last week of the Maintenance Treatment Period (Week 8) . If a patient's mean weekly pain score during the last week of the Maintenance Treatment Period is greater than the baseline score (i.e., the patient has an increase in pain compared to baseline), his/her response to treatment will be assigned a value of 0 (i.e. the patient will be considered a non-responder). Patients who discontinue study drug early will be considered non-responders to treatment and will be assigned a pain response of 0.
  The percentage of subjects achieving levels of treatment response 10% to 100% by 10% increments as defined above will be calculated with 30% of key interest as it has been shown to represent a clinically important improvement in pain.
Time Frame: Week 8
Measure: Number; unit: percentage of patients
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 316 | 160
percentage of patients | 41.5 | 50.6
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.1033, Regression, Logistic; Logistic regression, including treatment, baseline weekly pain score, and OA joint as independent variables; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.5 to 1.1] — Ratio between treatment odds of achieving a treatment response

7. Secondary Outcome: Proportion of Patients With at Least 50% Improvement From Baseline in the Weekly Mean Pain Intensity at Week 8
Description: as for outcome 6
Time Frame: Week 8
Measure: Number; unit: percentage of patients
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 316 | 160
percentage of patients | 25.6 | 31.3
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.2831, Regression, Logistic; Logistic regression, including treatment, baseline weekly pain score, and OA joint as independent variables; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.5 to 1.2] — Ratio between treatment odds of achieving a treatment response

8. Secondary Outcome: Proportion of Patients Whose OA Pain Was "Very Much Improved" or "Much Improved" as Indicated by Patient Global Impression of Change (PGIC) Score at Week 8
Description: The PGIC is a self-administered instrument that measures the patient's overall impression of his/her OA on a 7-point scale where 1 = "Very much improved" and 7 = "Very much worse".
Time Frame: Week 8
Measure: Number; unit: percentage of patients
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 316 | 160
percentage of patients | 44.3 | 40.0
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.1959, Regression, Logistic; Logistic regression with treatment as a main effect and OA joint as a covariate; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.9 to 2.0] — Ratio between treatment odds of having a PGIC of "Very Much Improved" or "Much Improved"

9. Secondary Outcome: Average Daily Number of Acetaminophen Tablets Used During Entire Study
Description: The average daily number of acetaminophen tablets used during the study will be calculated using data recorded in the patient diary as the sum of the total number of tablets used divided by the length of exposure (in days).
  The supplemental pain medication for OA will be grouped categorically into the following classes: (1) no supplemental acetaminophen tablets, (2) 0 to ≤ 0.5 tablets, (3) > 0.5 to ≤ 1.0 tablets, (4) > 1.0 to ≤ 2.0 tablets, and (5) > 2.0 tablets.
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: Tablets
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 316 | 160
Tablets | 0.5 (2.27) | 0.4 (1.75)
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.2858, Wilcoxon (Mann-Whitney); Wilcoxon Rank Sum test stratified by Primary OA joint (Hip or Knee) and Baseline Week Mean of the Daily NRS (<6.7 or >=6.7) (Van Elteren test)

10. Secondary Outcome: Proportion of Patients Withdrawing From Treatment Due to Lack of Analgesic Efficacy
Time Frame: Week 8
Measure: Number; unit: percentage of patients
Arm/Group | CR845 Tablet | Placebo Tablet
Number analyzed (Participants) | 316 | 160
percentage of patients | 2.5 | 3.1
Statistical Analysis 1: Comparison: CR845 Tablet vs Placebo Tablet; Test type: Superiority; p = 0.8002, Regression, Logistic; Logistic regression, including treatment, baseline pain score, and OA joint as independent variables; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.3 to 2.7] — Ratio between treatment odds of withdrawing from treatment due to lack of analgesic efficacy

ADVERSE EVENTS:
Time Frame: 59 Days
Description: Treatment emergent AEs (TEAEs) will be defined as AEs where onset occurs from the day of first dose of study medication up to and including the 2nd day following the day of last dose of study medication.
Arm/Group | CR845 Tablet | Placebo Tablet
All-Cause Mortality (participants affected / at risk) | 0/316 | 0/160
Serious Adverse Events (participants affected / at risk) | 9/316 | 1/160
Other Adverse Events (participants affected / at risk) | 82/316 | 17/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 Tablet (N=316) | Placebo Tablet (N=160)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 — Last Treatment Patient Received: CR845 2.5 mg
Cholecystitis (Hepatobiliary disorders) | 1 | 0 — Last Treatment Patient Received: CR845 1.0 mg
Pneumonia (Infections and infestations) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg; One patient experienced the serious adverse events of head injury, lumbar vertebral fracture, rib fracture, thoracic vertebral fracture, subdural haemorrhage and subarachnoid haemorhage.
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg; One patient experienced the serious adverse events of head injury, lumbar vertebral fracture, rib fracture, thoracic vertebral fracture, subdural haemorrhage and subarachnoid haemorhage.
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg; One patient experienced the serious adverse events of head injury, lumbar vertebral fracture, rib fracture, thoracic vertebral fracture, subdural haemorrhage and subarachnoid haemorhage.
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg; One patient experienced the serious adverse events of head injury, lumbar vertebral fracture, rib fracture, thoracic vertebral fracture, subdural haemorrhage and subarachnoid haemorhage.
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg; One patient experienced the serious adverse events of head injury, lumbar vertebral fracture, rib fracture, thoracic vertebral fracture, subdural haemorrhage and subarachnoid haemorhage.
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 — Last Treatment Patient Received: CR845 2.5 mg
Encephalopathy (Nervous system disorders) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg; One patient experienced the serious adverse events of head injury, lumbar vertebral fracture, rib fracture, thoracic vertebral fracture, subdural haemorrhage and subarachnoid haemorhage.
Mental Status Changes (Psychiatric disorders) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Last Treatment Patient Received: CR845 5.0 mg
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 Tablet (N=316) | Placebo Tablet (N=160)
Constipation (Gastrointestinal disorders) | 42 | 3
Dizziness (Nervous system disorders) | 26 | 3
Headache (Nervous system disorders) | 18 | 9
Dry mouth (Gastrointestinal disorders) | 18 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT02944448/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT02944448/SAP_001.pdf